CLINICAL TRIAL: NCT05370950
Title: A Single-center, Randomized, Parallel, Open-label Study to Compare the Bioavailability, Pharmacodynamics, and Safety of SHR-1209 Given as Single Subcutaneous Injection at Different Sites in Healthy Volunteers
Brief Title: Study of Bioavailability, Pharmacodynamics and Safety of SHR-1209 Administered by Single Subcutaneous Injection at Different Sites in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR-1209-104
Record Dates: First submitted 2022-05-07; First posted 2022-05-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Hypercholesterolemia and Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Single-center, random, parallel, open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1209
- Treatment group B (Experimental)
  Interventions: Drug: SHR-1209
- Treatment group C (Experimental)
  Interventions: Drug: SHR-1209

INTERVENTIONS:
Drug: SHR-1209 — SHR-1209，single subcutaneous injection of 450mg

SUMMARY:
In order to meet the preferences and needs of different patients for injection sites and improve the medication compliance of patients, it is planned to compare the bioavailability, pharmacokinetics, pharmacodynamic and safety data to assess feasibility of multiple injection sites for administration.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the research procedures and methods, being able to complete the research in accordance with the procedure requirements, and sign the informed consent;
2. The age on the date of signing the informed consent must be ≥18 years old and ≤55 years old;
3. Body mass index (BMI) at screening period must be ≥18.5 kg/m2 and <30.0 kg/m2, weight of male must≥ 50.0 kg and <90.0 kg, and female≥ 45.0 kg and <90.0 kg;
4. The subjects and their female partners are willing to have no reproductive plan from 2 weeks before screening to 6 months after the administration of the study drug, and voluntarily take effective contraceptive measures and do not plan to donate sperm or ovum.

Exclusion Criteria:

1. History of the following diseases or treatments:

   Diseases that affect drug absorption, distribution, metabolism, and excretion determined by the investigator; Serious infection within 3 months before screening; History of drug allergy or atopic allergic disease (asthma, urticaria).
2. Any one of the following tests at Screening period or Baseline period:

   Human immunodeficiency virus antibody (HIV-Ab), syphilis serological examination, hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab) positive; Positive blood pregnancy test.
3. General situation:

   Have a history of drug use or drug abuse; Women who are pregnant or breastfeeding.
4. Subjects who are considered by the investigator to have any other factors which are not suitable for participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: area under the curve (AUC0-t) | Days 1-113
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: area under the curve (AUC0-∞) | Days 1-113
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: peak concentration (Coax) | Days 1-113

SECONDARY OUTCOMES:
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: time to peak (Tmax) | Days 1-113
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: terminal elimination half-life (t1/2) | Days 1-113
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: apparent volume of distribution (Vz/F) | Days 1-113
Pharmacokinetic parameters of single subcutaneous injection of SHR-1209: apparent clearance (CL/F) | Days 1-113
Incidence and severity of adverse events (AE), serious adverse events (SAE), etc. | Days 1-113

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053
- [Derived] Wang Y, Cheng Y, Guo Y, Fan Y, Zhou R, Zhang Q, Xu Y, Feng S, Shen K, Hu W. A Phase I Study to Evaluate the Relative Bioavailability, Pharmacodynamics, and Safety of a Single Subcutaneous Injection of Recaticimab at Three Different Sites in Healthy Chinese Subjects. Eur J Drug Metab Pharmacokinet. 2025 May;50(3):265-272. doi: 10.1007/s13318-025-00944-5. Epub 2025 Apr 19. PMID 40252193